CLINICAL TRIAL: NCT05708612
Title: Safety and Performance of a Silicone Implant for Fecal Incontinence Treatment (SimplyFI)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: A.M.I. Agency for Medical Innovations GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CI-48-001; CIV-AT-23-01-041926 (Other: EUDAMED CIV-ID)
Record Dates: First submitted 2023-01-23; First posted 2023-02-01 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Fecal Incontinence
Keywords: Surgical Treatment; Implant
MeSH Terms: conditions — Fecal Incontinence | interventions — Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Implantation of SimplyFI (Experimental): Long-term non-active implant
  Interventions: Procedure: Medical Device (SimplyFI)

INTERVENTIONS:
Procedure: Medical Device (SimplyFI) — Implantation a non-active medical device (SimplyFI) for the treatment of chronic fecal incontinence.

SUMMARY:
The purpose of the clinical investigation is to verify that the device under investigation (SimplyFI) is appropriate to significantly improve fecal incontinence in patients in whom its use is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female subjects
* Age ≥ 18 years, <85 years
* Subject has failed standard conservative therapy for fecal incontinence (at least 6 months)
* Subject is a surgical candidate
* Subject is willing and able to cooperate with follow-up examinations
* Subject has been informed of the study procedures and the treatment and has signed an informed consent form and provided authorization to use and disclose information for research purposes.

Exclusion Criteria:

* Treatment with another investigational drug or investigational device
* Unable to understand study requirements or is unable to comply with follow-up schedule
* Contraindicated according to the instruction for use of the device
* Pregnancy or nursing, or plans to become pregnant
* History of significant obstructed defecation or other significant chronic defecatory motility disorders
* Current, external full thickness rectal prolapse or vaginal prolapse
* Inflammatory Bowel Disease
* Irritable Bowel Syndrome
* Systemic disease as source of FI (scleroderma, neurologic disorders, Crohn's)
* Active pelvic infection
* Chronic diarrhea
* Medical history of anal, rectal, or colon cancer
* Prior anterior resection of the rectum
* Medical history of pelvic radiation therapy
* Significant scarring of the recto-vaginal septum, a permanent implant in the rectovaginal septum, or a history of recto-vaginal fistula
* Previous anorectal posterior compartment surgery
* History of complex anal fistula

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Safety-related complications and adverse events | 12 months
  The primary endpoint is safety-related complications and adverse events during follow-up until 12 months after surgery.

SECONDARY OUTCOMES:
Cure of fecal incontinence (Fecal Incontinence Quality of Life Scale (FIQLs)) | 12 months
  The secondary endpoint is to evaluate the change of fecal incontinence assessed by validated scores (changes from baseline to 1 week, 1 months, 3 months, 6 months) until 12 months after surgery.
  Fecal Incontinence Quality of Life scale (all subscale scores 1-4). Scales range from 1 to 5, with a 1 indicating a lower functional status of quality of life. Scale scores are the average (mean) response to all items in the scale.
Quality of Life (St. Mark's incontinence score (SMIS)) | 12 months
  The secondary endpoint is to evaluate the change of Quality of Life assessed by validated scores (changes from baseline to 1 week, 1 months, 3 months, 6 months) until 12 months after surgery.
  St. Marks incontinence score contains 7 questions, and a higher total score means a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Riss, Prof. PD Dr., Principal Investigator — Medical University Vienna; José Manuel Devesa Múgica, Dr., Principal Investigator — Hospital Ruber Internacional
Locations (6):
- Austria (2):
  - Göttlicher Heiland Krankenhaus, Vienna
  - Medical University Vienna, Vienna
- Germany (2):
  - Klinikum Bielefeld Rosenhöhe, Bielefeld
  - MVZ Wiesbaden / KD Helios Klinik, Wiesbaden
- Spain (2):
  - Hospital Ruber Internacional, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dawoud C, Devesa JM, Lohnert M, Vicente R, Metwalli SA, Riss S. Artificial sphincter with a new silicone band for treating faecal incontinence: IDEAL 2b prospective multicentre trial. BJS Open. 2025 Sep 8;9(5):zraf112. doi: 10.1093/bjsopen/zraf112. PMID 41123163